CLINICAL TRIAL: NCT06521190
Title: Phase IIa Randomized, Double-blind, and Placebo-controlled Multicenter Split Body Trial of Repeated Doses of ACOU085 for the Prevention of Hearing Loss in Testicular Cancer Patients Receiving Cisplatin
Brief Title: ACOU085 for Hearing Loss Prevention in Testicular Cancer Patients Receiving Cisplatin
Acronym: PROHEAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acousia Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EUCT 2023-503696-15-00
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Cisplatin-induced Hearing Loss

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, and placebo-controlled multicenter split body trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active ear (Active Comparator): An ACOU085 retard formulation is transtympanically injected into the round window niche of the middle ear.
  Interventions: Drug: ACOU085 (bimokalner)
- Placebo ear (Placebo Comparator): A matching placebo retard formulation is transtympanically injected into the round window niche of the contralateral middle ear.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACOU085 (bimokalner) — Transtympanic injection
  Arms: Active ear
Drug: Placebo — Transtympanic injection
  Arms: Placebo ear

SUMMARY:
Randomized, double-blind, placebo-controlled, multicenter phase IIa clinical trial in adult male TCa patients with the risk to suffer from sensorineural hearing loss (SNHL) due to cisplatin therapy within a chemotherapeutic regimen of testicular cancer. Patients will have an indication for a cisplatin-containing chemotherapy according to current guidelines and trial site tumor board recommendations. The trial is designed to show efficacy, safety, and tolerability of ACOU085 administered into the middle ear using 3 transtympanic injections per ear prior to 3 planned and corresponding 3-week chemotherapeutic cycles. The intra-individual control will be done by placebo injection into the respective contralateral middle ear.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of testicular cancer with indication for a cis-Pt-containing chemotherapeutic regimen according to current treatment guidelines and site-specific tumor board recommendations
* Male adult patients at an age between 18 and 45 years
* Planned cis-Pt treatment with a cumulative dose of ≥300 mg/m2 which has to be administered in three chemotherapeutic cycles
* Normal or not clinically relevant otoscopic findings in both ears
* Normal hearing at both ears according to current WHO criteria for air-conduction 4PTA (0.5/1/2/4 kHz; 0 to 19 dB HL; average of audiometric thresholds at 0.5/1/2/4 kHz) at baseline
* Normal hearing at both ears according to ASHA criteria with a hearing threshold at any frequency (0.25 to 12 kHz) not exceeding 20 dB and a 4PTA (0.5/1/2/4 kHz) showing ≤15 dB HL at baseline
* Normal distortion product oto-acoustic emissions (DPOAE) present in both ears at baseline
* Patient shows normal results at trial start (V1) concerning heart rate (50 to 90 bpm), blood pressure (according to commonly accepted ranges), ECG (no pathological findings), and laboratory parameters (ie, liver and renal function values not clinically significant)
* Male patients and their female partner(s) must agree to use 2 forms of contraception (one of which must be a barrier method) during 6 months after trial start (V1)
* Patient is cooperative, able to understand all aspects of the trial, and able to speak German comparable to native speakers as per the investigator's discretion
* Patient has signed an approved informed consent form indicating that he understands the purpose of and procedures required for the trial, will follow the trial-specific measures, and is willing to participate in the trial

Exclusion Criteria:

* Suspected or diagnosed genetic predisposition to hearing loss (incl. DFNA2 rel. to KCNQ4)
* History of middle ear pathology or surgery, otitis externa, chronic otitis media, or recent acute otitis media (within ≤3 months)
* History of otologic surgery (excluding myringotomy tubes or simple tympanoplasty)
* Meniere's disease or secondary endolymphatic hydrops, auto immune hearing loss, inner ear pathology, fluctuating hearing loss, perilymph fistula, cochlear baro-trauma, radiation-induced hearing loss, retro-cochlear lesion, severe tympanosclerosis, atrophic tympanic membrane
* Hearing loss of >45 dB averaged at 6 and 8 kHz in either ear
* Sudden hearing loss or conductive hearing loss >10 dB at two frequencies in either ear
* Asymmetry in hearing thresholds between left and right ear ≥20 dB at any single frequency or ≥10 dB at any 3 consecutive frequencies ≤ 8 kHz
* Intake of any ototoxic drugs other than the intended cis-Pt-containing chemotherapeutic drug regimen prior to start of the trial and during the trial period
* Previous radiation exposure >35 Gray to complete or parts of the cochlea
* Severe concomitant diseases such as heart failure (NYHA II-IV), COPD, bronchial asthma, ongoing malignancies other than testicular cancer, auto-immune or chronic-inflammatory diseases, endocrinological diseases, advanced hepatic or renal failure, and primary complaint of tinnitus
* Planned consumption of medications, herbal preparations, and specific food ingredients to treat hearing problems and/or tinnitus during the trial period
* Hypersensitivity against any primary or secondary ingredient of IMP/Placebo medication
* Male patients with female partners who are pregnant or planning to become pregnant during 6 months after trial start (V1)
* Use of any other investigational medicinal product (IMP) within five times the half-life of that IMP/relevant metabolites or one month (whichever is longer) prior to screening and planned use during the trial or up to 30 days after trial completion
* Patient has any dependent relationship or employment status with respect to the trial site, the sponsor, the investigator, or any supervisor

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients with testicular cancer
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
PTA air | Visit 4 at 9 weeks
  Proportion of patients showing a difference of ≥10 dB between the ears in at least two frequencies for air conduction in PTA focused on high (4, 6, 8 kHz) and extended high frequencies (10, 12, 14, 16 kHz) between baseline (V1; prior to first initiation of cis-Pt-containing chemotherapy) and end of chemotherapeutic cycle 3 (V4)

SECONDARY OUTCOMES:
Distortion Product Otoacoustic Emissions (DPOAE) | 150 days
  Intraindividual differences between the ears at Visits 2-5
PTA bone | 150 days
  Intraindividual differences between the ears at Visits 2-5
Oldenburger Test (speech understanding) | 150 days
  Intraindividual differences between the ears at Visits 2-5
Freiburger Test | 150 days
  Intraindividual differences between the ears at Visits 2-5

CONTACTS AND LOCATIONS:
Overall Officials: Sven Becker, PD Dr., Principal Investigator — Dept. of Otolaryngology - Head and Neck Surgery, Tübingen University, Germany
Locations (10):
- Germany (10):
  - Dept. of Otolaryngology - Head and Neck Surgery, Tuebingen University, Tübingen, Baden-Wurttemberg
  - Dept. of Otolaryngology - Head and Neck Surgery, Dresden University, Dresden
  - Dept. of Otolaryngology - Head and Neck Surgery, Essen University, Essen
  - Department of Otolaryngology - Head and Neck Surgery, Hamburg University, Hamburg
  - Dept. of Otolaryngology - Head and Neck Surgery, Jena University, Jena
  - Dept. of Otolaryngology - Head and Neck Surgery, Mannheim University, Mannheim
  - Dept. of Otolaryngology - Head and Neck Surgery, Marburg University, Marburg
  - Dept. of Hematology and Oncology, Rotkreuzklinikum Munich, Munich
  - Dept. of Otolaryngology - Head and Neck Surgery, Munich Technical University, Munich
  - Dept. of Otolaryngology - Head and Neck Surgery, Wuerzburg University, Würzburg

IPD SHARING:
Plan to Share IPD: No